CLINICAL TRIAL: NCT06244615
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial of an Antiviral Mouth and Throat Rinse for the Treatment of Acute Sore Throat (Upper Respiratory Tract Infection e.g., Pharyngitis/Laryngitis)
Brief Title: Clinical Trial of a Mouth and Throat Rinse for the Treatment of Acute Sore Throat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Collaborators: Pharmaxi LLC (Industry); Labor Dr. Fenner und Kollegen (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LSMR-01/2022
Record Dates: First submitted 2023-12-19; First posted 2024-02-06 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Sore-throat; Upper Respiratory Infection
MeSH Terms: conditions — Pharyngitis; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Verum mouth and throat rinse (Experimental): Formulation containing WO 6607 for oral administration (rinse and gargle).
  Interventions: Device: Verum (WO 6607)
- Placebo mouth and throat rinse (Placebo Comparator): Formulation containing WO 6608 for oral administration (rinse and gargle).
  Interventions: Device: Placebo (WO 6608)

INTERVENTIONS:
Device: Verum (WO 6607) — Mouth and throat rinse and gargle solution
  Arms: Verum mouth and throat rinse
Device: Placebo (WO 6608) — Mouth and throat rinse and gargle solution
  Arms: Placebo mouth and throat rinse

SUMMARY:
The aim of this study is to confirm the efficacy, safety and tolerability of the Mouth and Throat Rinse in adult participants with acute sore throat (upper respiratory tract infection e.g., pharyngitis/laryngitis) compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having clinical signs and symptoms of recent (less than 48 h) acute sore throat (upper respiratory tract infection) without signs of lower respiratory tract infection (total severity score for throat irritation baseline value ≥ 4).
* Centor Score of 0 to 3 points at screening.
* Female and male subjects with 18-75 years of age.

Exclusion Criteria:

* Known allergy to any of the components in the investigational product (Placebo or Verum) (i.e. SLS).
* Centor Score of 4 points at screening.
* Presence of exanthema.
* Presence of oral mucosal plaques e.g., soor.
* Presence of bacterial infection of the upper respiratory tract (confirmed by rapid screening test).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Change in total severity score of throat irritation for subjective and objective symptoms during the clinical investigation (comparison between verum and placebo) | Day 1 vs Day 4
  A total severity score for throat irritation will be calculated at each visit as the sum of the subjective and objective symptoms. Each of the four criteria on a scale from 0 to 4:
  1. soreness, 2. difficulty swallowing (rated by the subject), 3. mucosal swelling of the throat and 4. oropharyngeal color (erythema) (assessed by the investigator)

SECONDARY OUTCOMES:
Evaluate the efficacy of the Verum Mouth and Throat Rinse compared to Placebo by analysing the detection of viruses | Day 1 vs. Day 2,Day 1 vs. Day 4, Day 1 vs. Day 7 and Day 1 vs. Day 14
  Combined nasal and oropharyngeal swab sampling for PCR detection of viruses including CT values reported for: Adenovirus, Coronaviruses including OC43, NL63, 229E and SARS-CoV-2, Influenza virus A and B, Parainfluenza virus 1-4, Rhinovirus, RSV) in adult subjects with acute sore throat (upper respiratory tract infection e.g., pharyngitis/laryngitis) compared to Placebo (Day 1 vs. Day 2 and Day 1 vs. Day 4)
Evaluate the efficacy of the Verum Mouth and Throat Rinse compared to Placebo with respect to the subjective symtoms of throat soreness and difficulty swallowing | Day 1 vs. Day 7±1 and Day 1 vs. Day 14±1
  Comparison between Verum and Placebo:
  Change Day 1 to Day 7±1 and Day 1 to Day 14±1 for each subjective symptom of throat soreness and difficulty swallowing (rated by the subject on a scale from 0 to 4)
Evaluate the efficacy of the Verum Mouth and Throat Rinse compared to Placebo regarding the objective symptoms of mucous swelling and oropharyngeal color (erythema) | Day 1 vs. Day 7±1 and Day 1 vs. Day 14±1
  Comparison between Verum and Placebo:
  Change Day 1 to Day 7±1 and Day 1 to Day 14±1 for each objective symptom of mucous swelling, oropharyngeal color (erythema) (assessed by the investigator on a scale from 0 to 4)
Evaluate the efficacy of the Verum Mouth and Throat Rinse compared to Placebo regarding the recovery time | Day 1 vs. Day 7 and Day 1 vs. Day 14
  Comparison between Verum and Placebo:
  Recovery time is defined as the time to improvement in total severity score of throat irritation value to ≤ 4, provided the score for each criterion is not > 1
Evaluate the efficacy of the Verum Mouth and Throat Rinse compared to Placebo regarding the proportion of rebound after treatment phase | Day 1 vs. Day 7 and Day 1 vs. Day 14
  Comparison between Verum and Placebo:
  Number of patients (%) with a rebound after treatment phase. Rebound is defined as worsening in total severity score of throat irritation value
Evaluate the efficacy of the Verum Mouth and Throat Rinse compared to Placebo regarding the proportion of expansion of the symptoms (e.g., subsequent bronchitis) | Day 1 vs. Day 7 and Day 1 vs. Day 14
  Comparison between Verum and Placebo:
  Number of patients in percent (%) having an expansion of the symptoms (e.g., subsequent bronchitis)
Evaluate the efficacy of the Verum Mouth and Throat Rinse compared to Placebo regarding the need for further medical intervention or treatments such as rescue therapy or pain medication | Day 1 vs. Day 7 and Day 1 vs. Day 14
  Comparison between Verum and Placebo:
  Number of patients with the need for further medical intervention or treatments such as rescue therapy or pain medication
Evaluate the efficacy of the Verum Mouth and Throat Rinse compared to Placebo regarding the presence of Metapneumovirus and Bocavirus | Day 1 vs. Day 4
  Comparison between Verum and Placebo:
  Combined nasal and oropharyngeal swab sampling for PCR detection of viruses without CT values reported for Metapneumovirus and Bocavirus
Global judgement of efficacy by the patient | Day 1 vs. Day 2, Day 1 vs. Day 7, Day 1 vs. Day 14
  The global judgement of efficacy (throat soreness and difficulty swallowing) will be assessed according to the severity score: 0= none, 1= mild, 2= moderate, 3= severe, 4= very severe
Global judgement of efficacy by the investigator | Day 1 vs. Day 2, Day 1 vs. Day 7, Day 1 vs. Day 14
  The global judgement of efficacy (mucous swelling and oropharyngeal color (erythema)) will be assessed according to the following scale: 0= none, 1= mild, 2= moderate, 3= severe, 4= very severe
Evaluate the safety of the Verum Mouth and Throat Rinse in adult subjects with acute sore throat (upper respiratory tract infection e.g., pharyngitis/laryngitis) | Day 1, Day 2, Day 3, Day 7±1, Day 14±1
  The safety will be assessed through adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Roman Fishchuk, MD, Principal Investigator — Central City Clinical Hospital of Ivano-Frankivsk
Locations (1):
- Central City Clinical Hospital of Ivano-Frankivsk, Ivano-Frankivsk, Ukraine